CLINICAL TRIAL: NCT06501417
Title: EC_ItaLynch: Incorporating Lynch Syndrome Genetic Testing in Standard Medical Care of Patients With Endometrial Cancer (Mainstreaming)
Brief Title: EC_ItaLynch: Mainstreaming the Diagnosis of Lynch Syndrome
Acronym: EC_ItaLynch
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6511
Record Dates: First submitted 2024-07-09; First posted 2024-07-15 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-04

CONDITIONS: Lynch Syndrome; Endometrial Cancer
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis; Endometrial Neoplasms | interventions — Gender Equity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: mainstreaming — mainstreaming in EC patients

SUMMARY:
Lynch syndrome (LS) is the most common cause of hereditary endometrial cancer (EC) and is associated with an increased risk of colorectal (CRC), ovarian, gastric, small bowel and urinary tract cancer. LS is determined by germline pathogenic variants in the DNA mismatch repair (MMR) genes (MLH1, MSH2, MSH6, PMS2) or in EPCAM.

Approximately 20-30% of ECs exhibit somatic MMR deficiency (dMMR), and among these patients approximately 10-30% are affected by LS. This estimate suggests that the prevalence of LS among all EC patients is roughly 3-5%. Prior to the introduction of Universal Screening, the diagnostic management of LS was mainly based on Selective Screening, which included clinical criteria based on the evaluation of family and personal history and the clinicopathological features of the tumor (Amsterdam criteria 1990, Bethesda criteria 1997). However, these have been limited in their application to clinical practice due to their complexity and the frequent lack of complete family history data. Therefore, Universal Screening for LS diagnosis by the identification of dMMR in the tumor tissue of all newly diagnosed CRC and EC cases has recently been proposed.

Universal Screening for LS in tumor tissue includes an immunohistochemistry based (IHC) test to assess loss of MMR protein expression or a polymerase chain reaction (PCR) test for microsatellite instability.

In the traditional diagnostic pathway for LS, genetic counseling and testing are always recommended for EC patients who are found to have loss of expression of any of the proteins encoded by the MSH2, MSH6, or PMS2. In case of MLH1 loss, genetic counseling and genetic testing are recommended for patients without hypermethylation of the MLH1 promoter.

Recent findings suggest that incorporating genetic testing in an oncologist-driven diagnostic algorithm (mainstreaming of genetic testing) could enable increased diagnostic rates, offering the benefits of precision medicine and a streamlined pathway of care to patients and their families.

The study consists of two parts:

1. In the first part the aim of the current study is to compare the knowledge, experience and understanding of genetic testing among patients pursuing genetic testing using mainstreaming or standard genetic counseling through modified Modified Royal Marsden Patient Satisfaction Questionnaire.
2. If the first aim will be achieved, a second part will be conducted, to evaluate the feasibility of the mainstreaming diagnostic pathway for LS.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of stage I-IV EC with dMMR
2. Only for part I presence of Lynch alert.
3. Signed Informed consent to participate in the study.
4. d. Patient must be ≥18 years

Exclusion Criteria:

1. Histologically confirmed diagnosis of stage I-IV EC with pMMR.
2. Significant psychiatric or clinical impairment compromising consent to the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: popolazione: sesso, anni, che accesso fanno, che patologia hanno..
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Patients satisfaction | 1 year
  The primary endpoint of this study is the rate of patients satisfied with the counseling measured by question n.15 of the Modified Royal Marsden Patient Satisfaction Questionnaire
LS diagnosis | 3 years
  the proportion of LS diagnosis in dMMR EC patients

CONTACTS AND LOCATIONS:
Overall Officials: Emanuela Lucci Cordisco, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy